CLINICAL TRIAL: NCT03016663
Title: LIPOFILLING IN BREAST SURGERY: VOLUMETRIC EVALUATION OF FAT RESORPTION AFTER WASHING WITH RINGER'S LACTATE
Brief Title: Volumetric Study of Fat Resorption After Breast Lipofilling
Acronym: Lipofilling
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: RP046D-15HTM
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Cosmetic Techniques; Mammaplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast Lipofilling Technique: Preliminary MRI breast were performed for volumetric measurement. Fat harvesting performed by same surgeon using water-assisted liposuction (WAL) and subsequent washing with buffered lactate in a standardized technique. Fat transfer performed using Berlin autologous lipotransplantation technique according to the BEAULI protocol .Patient were followed up monthly and MRI breast were repeated at 1st and 6th months after lipofilling. Clinical assessment and MRI Volumetric measurement performed using OsiriX (v7.0.3, 64 bit, Pixmeo c) software by same radiologist based on predefined operational procedure
  Interventions: Procedure: Technique of Breast Lipofilling

INTERVENTIONS:
Procedure: Technique of Breast Lipofilling — 1. Identification of the donor site Procedure carried out in single sessions under GA. Abdominal site identified and outlined with a skin marker.
  2. Fat Harvesting Berlin autologous lipotransplantation technique used according to the BEAULI protocol described by Ueberreiter et al.
     Infiltration solution -"Klein'solution" contains 1 cc of epinephrine (1:500,000) diluted in 500 cc of 0.001% lactate ringer solution (LRS).
  3. Fat Processing After aspiration of nonviable components of the aspirate, fat graft washed using Lactate Ringer Solution for three times. The fat processing and washing were performed by the same assistant for all patients.
  4. Fat Transfer (Injection) Fat is injected in small amounts as the needle is gradually withdrawn. Periglandular planes and intrapectoral planes are used. Intraparenchymal injection avoided.

SUMMARY:
Prospective observational study to evaluate effects on washing to improve viability of fat grafts in breast lipofilling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast defect post breast surgery and unsatisfied. The first lipofilling procedure delayed for at least 9 months after the completion of radiotherapy. Patient on chemotherapy deferred until at least 6 month of last chemotherapy.

Exclusion Criteria:

* Patients are excluded if they experienced local recurrence or distant metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with past history of breast cancer recruited.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measure fat graft resorption rate after washing with buffered lactate by volumeric MRI imaging | 6 month after breast lipofilling
  MRI Breast performed before the first lipofilling session, at 1st and 6th months after the lipofilling procedure. Volume measurement performed using OsiriX (v7.0.3, 64 bit , Pixmeo c)

SECONDARY OUTCOMES:
Confounding factors | 6 month after breast lipofilling
  To identify confounding factors that affect fat resorption rate in breast lipofilling To evaluate the fat resorption following breast lipofilling with volumetric MRI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Alizan ABDUL KHALIL, Principal Investigator — Department of Surgery University Malaya Medical Centre
Locations (1):
- University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiaschetti V, Pistolese CA, Fornari M, Liberto V, Cama V, Gentile P, Floris M, Floris R, Cervelli V, Simonetti G. Magnetic resonance imaging and ultrasound evaluation after breast autologous fat grafting combined with platelet-rich plasma. Plast Reconstr Surg. 2013 Oct;132(4):498e-509e. doi: 10.1097/PRS.0b013e3182a00e57. PMID 24076696
- [Background] Agha RA, Goodacre T, Orgill DP. Use of autologous fat grafting for reconstruction postmastectomy and breast conserving surgery: a systematic review protocol. BMJ Open. 2013 Oct 22;3(10):e003709. doi: 10.1136/bmjopen-2013-003709. PMID 24154518
- [Background] Petit JY, Lohsiriwat V, Clough KB, Sarfati I, Ihrai T, Rietjens M, Veronesi P, Rossetto F, Scevola A, Delay E. The oncologic outcome and immediate surgical complications of lipofilling in breast cancer patients: a multicenter study--Milan-Paris-Lyon experience of 646 lipofilling procedures. Plast Reconstr Surg. 2011 Aug;128(2):341-346. doi: 10.1097/PRS.0b013e31821e713c. PMID 21502905
- [Background] Claro F Jr, Figueiredo JC, Zampar AG, Pinto-Neto AM. Applicability and safety of autologous fat for reconstruction of the breast. Br J Surg. 2012 Jun;99(6):768-80. doi: 10.1002/bjs.8722. Epub 2012 Apr 4. PMID 22488516
- [Background] Sasaki GH. Water-assisted liposuction for body contouring and lipoharvesting: safety and efficacy in 41 consecutive patients. Aesthet Surg J. 2011 Jan;31(1):76-88. doi: 10.1177/1090820X10391465. PMID 21239675
- [Background] Ueberreiter K, von Finckenstein JG, Cromme F, Herold C, Tanzella U, Vogt PM. [BEAULI--a new and easy method for large-volume fat grafts]. Handchir Mikrochir Plast Chir. 2010 Dec;42(6):379-85. doi: 10.1055/s-0030-1267913. Epub 2010 Dec 15. German. PMID 21161858
- [Background] Crawford JL, Hubbard BA, Colbert SH, Puckett CL. Fine tuning lipoaspirate viability for fat grafting. Plast Reconstr Surg. 2010 Oct;126(4):1342-1348. doi: 10.1097/PRS.0b013e3181ea44a9. PMID 20885257
- [Background] Herold C, Knobloch K, Grimme M, Vogt PM. Does the injection plane matter in autologous fat transplantation? Aesthetic Plast Surg. 2010 Oct;34(5):678-9. doi: 10.1007/s00266-010-9490-1. No abstract available. PMID 20333518
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Kanchwala SK, Glatt BS, Conant EF, Bucky LP. Autologous fat grafting to the reconstructed breast: the management of acquired contour deformities. Plast Reconstr Surg. 2009 Aug;124(2):409-418. doi: 10.1097/PRS.0b013e3181aeeadd. PMID 19644255
- [Background] Hamza A, Lohsiriwat V, Rietjens M. Lipofilling in breast cancer surgery. Gland Surg. 2013 Feb;2(1):7-14. doi: 10.3978/j.issn.2227-684X.2013.02.03. PMID 25083450
- [Background] Saint-Cyr M, Rojas K, Colohan S, Brown S. The role of fat grafting in reconstructive and cosmetic breast surgery: a review of the literature. J Reconstr Microsurg. 2012 Feb;28(2):99-110. doi: 10.1055/s-0031-1287675. Epub 2011 Sep 16. PMID 21928171
- [Background] Losken A, Pinell XA, Sikoro K, Yezhelyev MV, Anderson E, Carlson GW. Autologous fat grafting in secondary breast reconstruction. Ann Plast Surg. 2011 May;66(5):518-22. doi: 10.1097/SAP.0b013e3181fe9334. PMID 21451387
- [Background] ELFadl D, Garimella V, Mahapatra TK, McManus PL, Drew PJ. Lipomodelling of the breast: a review. Breast. 2010 Jun;19(3):202-9. doi: 10.1016/j.breast.2010.02.009. Epub 2010 Mar 26. PMID 20347309
- [Background] Costantini M, Cipriani A, Belli P, Bufi E, Fubelli R, Visconti G, Salgarello M, Bonomo L. Radiological findings in mammary autologous fat injections: a multi-technique evaluation. Clin Radiol. 2013 Jan;68(1):27-33. doi: 10.1016/j.crad.2012.05.009. Epub 2012 Jun 30. PMID 22749812
- [Background] Shiffman MA, Mirrafati S. Fat transfer techniques: the effect of harvest and transfer methods on adipocyte viability and review of the literature. Dermatol Surg. 2001 Sep;27(9):819-26. doi: 10.1046/j.1524-4725.2001.01062.x. PMID 11553171
- [Background] Rennekampff HO, Reimers K, Gabka CJ, Germann G, Giunta RE, Knobloch K, Machens HG, Pallua N, Ueberreiter K, Heimburg Dv, Vogt PM. [Current perspective and limitations of autologous fat transplantation--"consensus meeting" of the German Society of Plastic, Reconstructive and Aesthetic Surgeons at Hannover; September 2009]. Handchir Mikrochir Plast Chir. 2010 Apr;42(2):137-42. doi: 10.1055/s-0030-1249672. Epub 2010 Mar 29. German. PMID 20352577
- [Background] Spear SL, Wilson HB, Lockwood MD. Fat injection to correct contour deformities in the reconstructed breast. Plast Reconstr Surg. 2005 Oct;116(5):1300-5. doi: 10.1097/01.prs.0000181509.67319.cf. PMID 16217471
- [Background] Smith P, Adams WP Jr, Lipschitz AH, Chau B, Sorokin E, Rohrich RJ, Brown SA. Autologous human fat grafting: effect of harvesting and preparation techniques on adipocyte graft survival. Plast Reconstr Surg. 2006 May;117(6):1836-44. doi: 10.1097/01.prs.0000218825.77014.78. PMID 16651956
- [Background] Schultz I, Lindegren A, Wickman M. Improved shape and consistency after lipofilling of the breast: patients' evaluation of the outcome. J Plast Surg Hand Surg. 2012 Apr;46(2):85-90. doi: 10.3109/2000656X.2011.653256. PMID 22471255
- [Background] Conde-Green A, de Amorim NF, Pitanguy I. Influence of decantation, washing and centrifugation on adipocyte and mesenchymal stem cell content of aspirated adipose tissue: a comparative study. J Plast Reconstr Aesthet Surg. 2010 Aug;63(8):1375-81. doi: 10.1016/j.bjps.2009.07.018. Epub 2009 Aug 12. PMID 19679523
- [Background] Hsu VM, Stransky CA, Bucky LP, Percec I. Fat grafting's past, present, and future: why adipose tissue is emerging as a critical link to the advancement of regenerative medicine. Aesthet Surg J. 2012 Sep;32(7):892-9. doi: 10.1177/1090820X12455658. PMID 22942117
- [Background] Mestak O, Hromadkova V, Fajfrova M, Molitor M, Mestak J. Evaluation of Oncological Safety of Fat Grafting After Breast-Conserving Therapy: A Prospective Study. Ann Surg Oncol. 2016 Mar;23(3):776-81. doi: 10.1245/s10434-015-4908-2. Epub 2015 Oct 14. PMID 26467459
- [Background] Uda H, Sugawara Y, Sarukawa S, Sunaga A. Brava and autologous fat grafting for breast reconstruction after cancer surgery. Plast Reconstr Surg. 2014 Feb;133(2):203-213. doi: 10.1097/01.prs.0000437256.78327.12. PMID 24150122